CLINICAL TRIAL: NCT07165067
Title: A Phase 1, Open-label Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Activity of AP601 in Patients With Solid Tumors.
Brief Title: A Study of AP601 in Patients With Locally Unresectable Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AP Biosciences Inc. (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AP601-101
Record Dates: First submitted 2025-08-20; First posted 2025-09-10 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumours
Keywords: solid tumours; advanced or metastatic solid tumours; open label

STUDY DESIGN:
Intervention Model Description: AP601 is a fully human bispecific antibody designed for the treatment of CD73-expressing solid tumours. AP601 represents an innovative therapeutic approach, targeting both CD73 and CD137 to synergistically enhance antitumour immunity through two synergistic mechanisms. CD73, an ecto-enzyme frequently overexpressed in various cancers, plays a pivotal role in immune suppression by converting adenosine monophosphate into adenosine, which suppresses T cell activity within the tumour microenvironment (TME). By inhibiting CD73, AP601 mitigates adenosine-mediated immunosuppression, fostering a more effective immune response. Simultaneously, AP601 targets CD137, a key costimulatory receptor on activated T cells and natural killer cells. Engagement of CD137 stimulates proliferation and enhances the cytotoxic function of these immune cells. AP601's dual-targeting design restricts CD137 activation to the TME. This targeted approach minimizes systemic toxicity and enhances therapeutic specificity.
Masking Description: Open Label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Cohort 1: 0.5 mg/kg Participants will receive a single infusion of AP601 once every 2 weeks (14 days)
  Interventions: Drug: AP601
- Cohort 2 (Experimental): Cohort 2: 1.25 mg/kg Participants will receive a single infusion of AP601 once every 2 weeks (14 days)
  Interventions: Drug: AP601
- Cohort 3 (Experimental): Cohort 3: 2.5 mg/kg Participants will receive a single infusion of AP601 once every 2 weeks (14 days)
  Interventions: Drug: AP601
- Cohort 4 (Experimental): Cohort 4: 5.0 mg/kg Participants will receive a single infusion of AP601 once every 2 weeks (14 days)
  Interventions: Drug: AP601
- Cohort 5 (Experimental): Cohort 5: 7.5 mg/kg
  Interventions: Drug: AP601
- Cohort 6 (Experimental): Cohort 6: 10.0 mg/kg
  Interventions: Drug: AP601

INTERVENTIONS:
Drug: AP601 — AP601 is a fully human bispecific antibody designed for the treatment of CD73-expressing solid tumours. Participants will receive a single infusion of AP601 once every 2 weeks (14 days) (Q2W) for up to 12 months. All doses of AP601 will be admistered intraveneously. The infusion time for all doses of AP601 in each patient will be approximately 60 to 120 minutes.

SUMMARY:
A Phase 1, Open-Label Study of the Safety, Tolerability,Pharmacokinetics, Pharmacodynamics and Clinical Activity of AP601 in Patients with Solid Tumours.The study is designed to find the highest dose of AP601 that can be given safely. Participants will be assigned to one of six cohorts. Each cohort will receive a different dose of the study medication, AP601, based on the body weight. Each cohort will initially enrol 1-3 participants. If no serious side effects are seen in the first participant(s), the next cohort will receive the next dose level.

DETAILED DESCRIPTION:
Participants will receive a single infusion of AP601 once every 2 weeks (14 days) (Q2W) for up to 12 months.

Part 1 (Dose Escalation):

Part 1 is a dose escalation part, using an accelerated 3+3 design. Up to 6 dose levels are planned to be evaluated in Part 1.

Cohort 1 - 0.5mg/kg (1-6 participants) Cohort 2 - 1.25 mg/Kg (1-6 participants) Cohort 3 - 2.5 mg/Kg (3-6 participants) Cohort 4- 5.0 mg/Kg (3-6 participants) Cohort 5- 7.5 mg/Kg (3-6 participants) Cohort 6- 10.0 mg/Kg. (3-6 participants) At the first dose level, a single participant will be enrolled and observed for dose-limiting toxicities (DLTs) and adverse events (AEs) for 28 days (2 treatment cycles). If the participant does not experience any DLTs, then a new participant may be dosed at the next higher dose level and observed for the DLT period (28 days). There will be a maximum of 2 single-patient cohorts.

If in any of the single-patient cohorts a patient experiences a DLT, an additional 2 patients will be enrolled at that dose level and evaluated using 3+3 design rules.

Cohorts 3 and above will all use a standard 3+3 design, even if toxicity was not seen in the single-patient Cohorts 1 and 2.

Part 2 (Dose Expansion):

A dose expansion part may be initiated following completion of the dose escalation cohorts.

ELIGIBILITY:
Inclusion Criteria: 1. Patients with histologically or cytologically proven locally unresectable advanced or metastatic solid tumors. Patients must be relapsed or refractory to at least one standard-of-care therapy, and/or have refused standard-of-care therapy.

2. Eastern Cooperative Oncology Group performance status of 0 to 1 at Screening, with an estimated life expectancy of at least 3 months.

3. Disease must have at least 1 assessable (long diameter ≥1 cm) lesion for evaluation of response by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

4. Patients with adequate organ and bone marrow function, in the absence of growth factors, including the specific laboratory findings of Absolute neutophil count, platelet count, Haemoglobin, AST, ALT, Serum total Bilirubin, Alkaline phosphatase, prothrombin time, INR or activated partial thromboplastin time, creatinine and albumin.

5. Female Volunteers must be of nonchild bearing potential i.e, surgically sterilised at least 6 weeks before Screening Visit or postmenopausal.

6. Females of childbearing potential must have a negative pregnancy test, agree not to attempt to become pregnant or donate Ova and agree to use contraception from one month prior to Screening until at least 90 days after last dose of study drug, if not exclusively in a same-sex relationship or abstinent as a committed lifestyle.

Male Vonuteers:

* Must agree not to donate sperm from signing the ICF until at aleast 90 days after the last dose of the study drug.
* If engaging in sexual intercourse with a female partner who could become pregnant, must agree to use adequate contraception.
* Willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. Has received concurrent antitumor treatment or IPs within 28 days of C1D1. The antitumor treatments include chemotherapy, radiotherapy, immunotherapy, targeted therapy, hormonal therapy, or cytokine therapy.
2. Has received prior CD73-targeted and/or CD137-targeted therapeutics.
3. Has had major surgery within 28 days prior to C1D1 (excluding prior diagnostic biopsy).
4. Any unresolved toxicity (except alopecia) from prior therapy of ≥CTCAE Grade 1, prior to the day of the first dose of IP. Participants with Grade 2 toxicity that is not CS (e.g., alopecia, vitiligo), or that is deemed stable or irreversible (e.g., peripheral neuropathy) can be enrolled.
5. History of any other malignancy, which has been active or treated within the past 2 years, with the exception of thyroid cancer, cervical intraepithelial neoplasia, basal cell carcinoma and squamous cell carcinoma.
6. Prior history of an irAE with immunotherapy-related toxicities that resulted in discontinuation of prior immunotherapy.
7. Current symptomatic leptomeningeal disease or uncontrolled, untreated brain metastasis.
8. Has received any organ transplantation including allogeneic stem cell transplantation.
9. Has received blood transfusions or growth factor support ≤ 14 days prior to screening.
10. Has any significant acute or chronic infections including:

    1. Infection requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days before first dose of AP601.
    2. Known active hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.
11. Current active, or history of, any autoimmune disease that may relapse or immunodeficiencies.
12. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before first dose of AP601.
13. Known severe hypersensitivity reactions to monoclonal antibodies.
14. Breastfeeding (or planning to breastfeed) at any time during the study, and for 90 days following study completion.
15. Participants with a current or recent (within the past 12 months) diagnosis of alcohol or non-prescribed drug abuse, as defined by local guidelines.
16. Evidence of cardiac dysfunction (defined as myocardial infarction within the last 6 months, New York Heart Association Class II/III/IV heart failure, unstable angina, unstable cardiac arrhythmias, or known left ventricular ejection fraction [LVEF] <55%) or other CS cardiac pathology likely to impair the participants ability to participate in the study.
17. Uncontrolled intercurrent illness including, but not limited to, uncontrolled hypertension, uncontrolled diabetes, uncontrolled endocrinopathy, severe active peptic ulcer disease or gastritis.
18. Has received a live (or live attenuated) vaccination within 28 days of the first dose of AP601 and during the study period.
19. Any other condition or prior therapy that in the opinion of the PI (or delegate) would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2027-12-27 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
To determine the tolerability (MTD and/or maximum administered dose [MAD] of AP601 in patients with solid tumours. | Initial 28 days from the first dose of AP601 which is Cycle1Day1 (each cycle is 14 days) until Cycle2Day14 (each cycle is 14 days)
  Estimate of the MTD based on DLTs observed during the DLT evaluation period.
To determine the tolerability of Recommend Phase 2 Dose [RP2D])- MTD and/or maximum administered dose [MAD] of AP601 in patients with solid tumours. | TEAEs and SAEs will be assessed at Screening until 90-day safety follow up visit.
  RP2D is based on the safety data - Estimate of the MTD based on DLTs observed during the DLT evaluation period
To determine the tolerability of Recommend Phase 2 Dose [RP2D]) | Cycle 1 - pre-dose, immediately following End of Infusion (EOI), 4 hours, 24 hours, 72 hours, 168 hours. Cycle 2- pre-dose, EOI, 4 hours, 24hours, 72hours, 168hours, Cycle 3 to Cycle 24- Predose (each cycle is 14 days), 0-6 hours, End of Trial Visit.
  RP2D tolerability is based on Pharmacokinetics data- blood samples will be collected to assess this.
To determine the tolerability of Recommend Phase 2 Dose [RP2D]) | PD will be assessed Cycle 1 - pre-dose, 24 hous, 72 hours, 168 hours. Cycle 2- pre-dose, 4 hours, 24hours, 72hours, 168hours, Cycle 3 to Cycle 24- Pre-dose (each cycle is 14days) and at End of Trial Visit.
  RP2D tolerability is based on Pharmacodynamics data- blood samples will be collected to assess this
To determine the tolerability of Recommend Phase 2 Dose [RP2D] | Antitumour activity data will collected at End of Trial Visit , Safety Follow Up Visit (End of Trial + 30 days), Safety FUP Visit (End of Trial + 90 days) and at Survival Follow Up.
  Recommend Phase 2 Dose [RP2D] is based on antitumor activity data.
To determine the tolerability of RP2D - Number of Participants with a Change from baseline in clinical laboratory parameters (haematology) | Assessed at Screening, Cycle1 Day1 , Cycle2 Day1, Cycle 3 Day1 to Cycle 24 Day 1(each cycle is of 14 days), End of Trial Visit (EOT) and Safety Follow Up (EOT+ 30 days)
  Haematology - blood samples will be collected. All safety laboratory assessments will be assessed by a local laboratory according to their reference ranges.
To determine the tolerability of RP2D - Number of Participants with a Change from baseline in clinical laboratory parameters (clinical chemistry) | Assessed at Screening, Cycle1 Day1 , Cycle2 Day1, Cycle3 Day1 until Cycle 24 Day 1 (each cycle is of 14 days), End of Trial Visit and Safety FUP (EOT+ 30 days)
  Clinical Chemistry- blood samples will be collected. All safety laboratory assessments will be assessed by a local laboratory according to their reference ranges.
To determine the tolerability of RP2D - Number of Participants with a Change from baseline in clinical laboratory parameters (Coagulation) | Assessed at Screening, Cycle1 Day1 , Cycle2 Day1, Cycle3 Day1 to last Cycle 24 Day 1(each cycle is of 14 days), End of Trial Visit and Safety FUP (EOT+ 30 days)
  Coagulation- blood samples will be collected. All safety laboratory assessments will be assessed by a local laboratory according to their reference ranges.
To determine the tolerability of RP2D - Number of Participants with a Change from baseline in clinical laboratory parameters (Thyroid Function tests ) | Assessed at Screening, Cycle1 Day1 , Cycle2 Day1, Cycle3 Day1 - until last Cycle 24 Day 1 (each cycle is of 14 days), End of Trial Visit and Safety FUP (EOT+ 30 days)
  Thyroid Function tests - blood samples will be collected. All safety laboratory assessments will be assessed by a local laboratory according to their reference ranges.
To determine the tolerability of RP2D - Number of Participants with a Change from baseline in clinical laboratory parameters (urinalysis) | Assessed at Screening, Cycle1 Day1 , Cycle2 Day1, Cycle3 Day1 - until last Cycle 24 Day 1 (each cycle is of 14 days), End of Trial Visit and Safety FUP (End of Trial Visit+ 30 days)
  Urine samples will be collected. All safety laboratory assessments will be assessed by a local laboratory according to their reference ranges.
To determine the tolerability of RP2D - Number of Participants with a Change from baseline in Vital signs measurements Pulse rate [PR], systolic and diastolic blood pressure [BP], temperature and respiratory rate [RR] | Assessed at Screening, Cycles 1 and 2 - Day 1, Day 2, Day 4, Day 8 Cycle 3 Day 1 - until last cycle 24 Day 1 (each cycle is 14 days), End of Trial Visit (EOT), Safety FUP (EOT + 30 days).
  Blood pressure will be measured using a sphygmomanometer, body temperature will be measured using a thermometer, Heart rate (HR) is measured using vital sign machine, respiratory rate is measured manually via 60-second count [RR]. All abnormal assessments measured as Clinically significant post dose will be recorded as AEs.
To determine the tolerability of RP2D- Number of Participants with a Change from baseline in body weight | Assessed at Screening, Cycles 1 and 2 - Day 1, Day 2, Day 4, Day 8 Cycle 3 Day 1 - until last cycle 24 Day 1(each cycle is 14 days), End of Trial Visit(EOT), Safety FUP (EOT + 30 days).
  Weight will be measured utilising scales.
To determine the tolerability of RP2D- Change from baseline in Eastern Cooperative Oncology Group (ECOG) score | Assessed at Screening, Cycle1 Day1, Cycle2 Day1, Cycle3 Day1 up until last cycle 24 Day1 (each cycle is of 14 days), End of Trial Visit(EOT)and Safety FUP (EOT + 30 days) Visit.
  Graded using a 6 point scale
To determine the tolerability of RP2D- Change from baseline in measurements of HR in beats per minute | Assessed at Screening, Cycle1 Day1, Cycle2 Day1, Cycle3 Day1 until last cycle 24 Day 1(each cycle is of 14 days), End of Trial Visit(EOT) and Safety FUP (EOT + 30 days).
  12-lead ECG parameters include the measurements of HR in beats per minute. All ECGs will be performed in triplicate.
To determine the tolerability of RP2D- Change from baseline in measurements of PR interval via 12-lead electrocardiogram | Assessed at Screening, Cycle1 Day1, Cycle2 Day1, Cycle3 Day1 until last cycle 24 Day 1(each cycle is of 14 days), End of Trial (EOT ) Visit and Safety FUP (EOT + 30 days).
  12-lead ECG parameters include the measurements of PR interval. All ECGs will be performed in triplicate.
To determine the tolerability of RP2D- Change from baseline in measurements of QT interval via 12-lead electrocardiogram | Assessed at Screening, Cycle1 Day1, Cycle2 Day1, Cycle3 Day1 until last cycle 24 Day 1(each cycle is of 14 days), End of Trial (EOT) Visit and Safety FUP (EOT + 30 days).
  12-lead ECG parameters include measurements of QT duration. All ECGs will be in triplicate.
To determine the tolerability of RP2D- Change from baseline in measurements of QRS duration via 12-lead electrocardiogram | Assessed at Screening, Cycle1 Day1, Cycle2 Day1, Cycle3 Day1 until last cycle 24 Day 1(each cycle is of 14 days), End of Trial (EOT) Visit and Safety FUP (EOT + 30 days).
  12-lead ECG parameters include the measurements of QRS duration. All 12-lead ECGs will be in triplicate.

SECONDARY OUTCOMES:
To assess the PK of AP601 in patients with solid tumours - Serum PK concentration of AP601. | Cycle 1 - Pre-dose, immediately following End of Infusion (EOI), 4 hours, 24 hours, 72 hours, 168 hours. Cycle 2- pre-dose, EOI, 4 hours, 24hours, 72hours, 168hours, Cycle 3 to Cycle 24 - Predose (each cycle is 14 days), 0-6 hours and End of Trial Visit.
  Blood samples will be collected to assess PK.
To assess the PK of AP601 in patients with solid tumours - Individual maximum concentration values, directly determined from the serum concentration time profiles for each participant (Cmax) | Cycle 1 - pre-dose, immediately following End of Infusion (EOI), 4 hours, 24 hours, 72 hours, 168 hours. Cycle 2- pre-dose, EOI, 4 hours, 24hours, 72hours, 168hours, Cycle 3 to Cyle 24- Predose(each cycle is 14 days), 0-6 hours and End of Trial Visit.
  Blood samples are collected to assess PK.
To assess the PK of AP601 in patients with solid tumours -Serum clearance following IV administration (CL) | Cycle 1 - Pre-dose, immediately following End of Infusion (EOI), 4 hours, 24 hours, 72 hours, 168 hours. Cycle 2- pre-dose, EOI, 4 hours, 24hours, 72hours, 168hours, Cycle 3 -to Cycle 24- Predose(each cycle is 14days), 0-6 hours and End of Trial Visit.
  Blood samples are collected to assess PK.
To assess the PK of AP601 in patients with solid tumours -Area under the serum concentration-time curve (AUC) from time zero to 168 hours post-dose (AUC0-168) | Cycle 1 - Pre-dose, immediately following End of Infusion (EOI), 4 hours, 24 hours, 72 hours, 168 hours. Cycle 2- pre-dose, EOI, 4 hours, 24hours, 72hours, 168hours, Cycle 3 to Cycle 24 Predose(each cycle is 14days), 0-6 hours and End of Trial Visit.
  Blood samples are collected to assess PK.
To assess the PK of AP601 in patients with solid tumours - AUC from time zero to the last time point with measurable concentration using the linear trapezoidal rule (AUClast) | Cycle 1 - Pre-dose, immediately following End of Infusion (EOI), 4 hours, 24hours, 72 hours, 168 hours. Cycle 2- pre-dose, EOI, 4 hours, 24hours, 72hours, 168hours, Cycle 3 to Cycle 24- Predose(each cycle is 14days), 0-6 hours and End of Trial Visit.
  Blood samples are collected to assess PK.
To assess the PK of AP601 in patients with solid tumours - The time to attain maximum concentration (Tmax) | Cycle 1 - pre-dose, immediately following End of Infusion (EOI), 4 hours, 24 hours, 72 hours, 168 hours. Cycle 2- pre-dose, EOI, 4 hours, 24hours, 72hours, 168hours, Cycle 3 to Cycle 24- Predose (each cycle is 14days), 0-6 hours and End of Trial Visit.
  Blood samples are collected to assess PK.
To assess the PK of AP601 in patients with solid tumours - Terminal elimination half-life (T1/2) | Cycle 1 - Pre-dose, immediately following End of Infusion (EOI), 4 hours, 24 hours, 72 hours, 168 hours. Cycle 2- pre-dose, EOI, 4 hours, 24hours, 72hours, 168hours, Cycle 3 to Cycle 24- Predose(each cycle is 14days), 0-6 hours and End of Trial Visit.
  Blood samples are collected to assess PK.
To assess the PK of AP601 in patients with solid tumours - Volume of distribution (Vz) | Cycle 1 - pre-dose, immediately following End of Infusion (EOI), 4 hours, 24 hours, 72 hours, 168 hours. Cycle 2- pre-dose, EOI, 4 hours, 24hours, 72hours, 168hours, Cycle 3 to Cycle 24- Predose(each cycle is 14days), 0-6 hours and End of Trial Visit.
  Blood samples are collected to assess PK.
To assess the PK of AP601 in patients with solid tumours - Trough concentration (Ctrough) | Cycle 1 - pre-dose, immediately following End of Infusion (EOI), 4 hours, 24 hours, 72 hrs, 168 hours. Cycle 2- pre-dose, EOI, 4 hours, 24hours, 72hours, 168hours, Cycle 3 to Cycle 24- Predose(each cycle is 14days), 0-6 hours and End of Trial Visit.
  Blood samples are collected to assess PK.
To assess the Immunogenicity of AP601 in patients with solid tumours. | Assessed at Cycle1 Day1 - Pre-dose, Cycle2 Day1 - Predose, Cycle3 Day1- Predose until Last Cycle 24 Day 1 (each cycle is of 14 days) and End of Trial Visit.
  Immunogenicity parameters will be assessed through analysis of the number and percentage of patients who develop anti-drug antibodies (ADA).
To assess the antitumor activity of AP601 in patients with solid tumours. | Antitumour activity data will collected at End of Trial(EOT) Visit , Safety FUP Visit (EOT + 30 days), Safety Follow Up Visit (EOT + 90 days) and at Survival Follow Up.
  This data will be collected through a follow up phone call following the last dose of AP601, through to last contact with the participant.
To evaluate the preliminary efficacy of AP601 in patients with solid tumours- Objective Response Rate (ORR) | Upto 2 years
  Preliminary efficacy will be assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
To evaluate the preliminary efficacy of AP601 in patients with solid tumours- Disease Control Rate (DCR) | Upto 2 years
  Preliminary efficacy will be assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
To evaluate the preliminary efficacy of AP601 in patients with solid tumours- Clinical Benefit Response (CBR) | Upto 2 years
  Preliminary efficacy will be assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Pindara Private Hospital, Brisbane, Queensland
  - Epworth HealthCare, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
Our IPD sharing plan is not yet developed. We will consider data sharing at a later date.